CLINICAL TRIAL: NCT04695626
Title: Prospective Randomized Controled Study on the Outcome of Greenhouse Tec in the Arthroscopic Treatment of Small and Medium Rotator Cuff Tear
Brief Title: Prospective Randomized Controled Study on the Outcome of Greenhouse Tec in the Arthroscopic Treatment of Small to Medium Rotator Cuff Tear
Status: Completed | Type: Observational
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Other Study IDs: GY
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Bone Marrow Stimulating; Modified Suture Bridge
Keywords: Rotator Cuff Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Greenhouse Group: The patients in this group will be underwent Greenhouse tec to repair tendon tears.
  Interventions: Procedure: The combination of bone marrow stimulation and modified suture bridge(Greenhouse tec)
- Traditional Single Row Group: The patients in this group will be underwent traditional single row repair to repair tendon tears.

INTERVENTIONS:
Procedure: The combination of bone marrow stimulation and modified suture bridge(Greenhouse tec) — According to the anteroposterior diameter of the injury, single or double high braided thread were used to suture the tendon in a modified Mason Allen way without knotting. Bone marrow stimulation was carried out in the footprint area of rotator cuff. A 2.0 mm diameter cone was created with a depth of 1 cm and a spacing of 5 mm. Six to eight holes were made due to the diameter of the tear of rotator cuff until blood and fat droplets exudate. Then the threads were passed through the locking eyelet of the lateral row anchor. After tightening the threads, the anchor was screwed in at the distal part of the gteater tuberosity. With this new technique, the rotator cuff was repaired by one lateral row anchor without medial row knotting.
  Groups: Greenhouse Group

SUMMARY:
This study is aprospective cohort study on the outcome of a combination of bone marrow stimulation and modified suture bridge in the arthroscopic treatment of small and medium rotator cuff tear. The patients with small to medium rotator cuff injuries (less than 3cm in diameter) requiring arthroscopic surgery were collected. The patients were followed up before and 6 weeks, 3 months, 6 months and 12 months after surgery, including pain, functional score, joint range of motion, MRI and CT findings, complications and other quantitative and qualitative indicators. The self-control and intra group analysis were performed to evaluate the treatment effect; and the correlation analysis was performed on the treatment results To determine the important factors affecting the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopy confirmed small to medium rotator cuff injury
* The data of preoperative functional examination were complete
* Unilateral rotator cuff injury
* Clinical follow-up can be completed

Exclusion Criteria:

* Anterior superior rotator cuff injury with simple subscapular injury or combined subscapular injury
* Previous shoulder surgery (incision or arthroscopy)
* Combined with diseases of other parts of the same limb
* Combined with Bankart injury, acromioclavicular joint disease, greater tuberosity fracture, glenoid fracture and so on
* Bilateral onset
* Unable or unwilling to receive clinical follow-up

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: According to the inclusion and exclusion criteria, 40 patients with small to middle rotator cuff injury treated by this technique（Greenhouse tec） in our hospital from September 2020 to December 2021 were included.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons'Form，ASES score | 1 year postoperatively
  A score used to evaluated the shoulder function

SECONDARY OUTCOMES:
Integrity of the tendon in MRI | 1 year postoperatively
  MRI was performed to identify the status of the tendon

OTHER OUTCOMES:
the condition of bone healing in CT | 1 year postoperatively
  CT was performed to identify the status of the bone healing

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China